CLINICAL TRIAL: NCT02448849
Title: Use of Autologous Bone Marrow Derived Mesenchymal Stromal Cells in Combination With Platelet Lysate Product for Human Long Bone Nonunion Treatment, A Phase 2-3 Clinical Trial
Brief Title: Autologous BM-MSC Transplantation in Combination With Platelet Lysate (PL) for Nonunion Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Bone-013
Record Dates: First submitted 2015-05-05; First posted 2015-05-20 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-09

CONDITIONS: Bone Fracture
Keywords: Autologous; nonunion fracture; bone marrow; mesenchymal; stromal cell; platelet lysate product
MeSH Terms: conditions — Fractures, Bone; Fractures, Ununited | interventions — Administration, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSC recipients (Experimental): The patients with nonunion fracture who underwent percutaneous implantation of bone marrow derived mesenchymal stem cells in combination with platelet lysate product.
  Interventions: Biological: Percutaneous injection
- Placebo (Placebo Comparator): The patients with nonunion fracture who underwent percutaneous injection of placebo.
  Interventions: Other: Percutaneous injection

INTERVENTIONS:
Biological: Percutaneous injection — percutanous implantation of bone marrow derived mesenchymal stromal cells in patients with nonunion fracture.
  Arms: MSC recipients
Other: Percutaneous injection — Percutaneous implantation of placebo in patients with nonunion fracture.
  Arms: Placebo

SUMMARY:
Nonunion of long bones would occur in almost 10% of fractures and because of its long term and complicated treatment, is known as a therapeutic challenge for both of the surgeons and patients.

Cell therapy is useful in treatment of nonunion and mesenchymal stromal/stem cells are the best candidates for this kind of treatment.

Percutaneous implantation of autologous bone marrow derived mesenchymal stromal/stem cell in combination with PL will be done in 30 patients with tibia nonunion. The other 30 patients as the control group will receive placebo. The patients will be followed at 2weeks, 3months, 6m and 12 months after implantation.

The Spss(v16) software will be used for data analysis.

DETAILED DESCRIPTION:
Long bone nonunion is known as a therapeutic challenge for both the orthopedic surgeons and the society. Current treatment of this disorder is autologous bone graft. This treatment has potential minor and major complications and is considered as a risky treatment. So researches are focused on new treatment approaches for this disease.

Cell therapy is one of these new approaches especially based on mesenchymal stromal cells.

The investigators will evaluate safety and efficacy of percutaneous implantation of autologous BM-MSC (bone marrow -derived mesenchymal stromal cell) in combination with PL (platelet lysate product) in 30 tibia nonunion patients. The other 30 patients will receive placebo. These patients will be followed up and data will be analyzed with spss(v16).

ELIGIBILITY:
inclusion criteria:

* Non-united fracture of tibial midshaft at X-ray.
* Non-united gap less than 1cm.
* Fracture has fixed by closed intramedullary rod.
* Hypotrophic type.
* At least 6 months after initial surgery.
* Patient informed consent.

Exclusion criteria:

* Infected nonunion
* Multiple major fracture
* Non treated major fracture
* malignancy
* Pregnancy or lactating
* Uncontrolled chronic diseases, such as: diabetes mellitus, hypertension, renal diseases, liver diseases, thyroid diseases, heart diseases, blood diseases, etc.
* Steroid usage.
* Positive test for HIV and/or HBS and/or HBC and/or HTLV (1,2)
* Fracture site more than 1 cm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
clinical union | 3months
  - Clinical union is defined as an asymptomatic patient who was able to fully bear weight on the injured leg
Radiological healing | 1week
  - radiographic fracture healing is defined by bone continuity (bony bridging) present in three out of four cortices in two projections (anterior-posterior & lateral x-rays), assessed by a blinded senior orthopedic surgeon.
  CT scan, for confirm the results - radiolographic fracture healing is defined by bone continuity (bony bridging) present in three out of four cortices in two projections (anterior-posterior & lateral x-rays), assessed by a blinded senior orthopedic surgeon.
  CT scan, for confirm the results
  - radiolographic fracture healing is defined by bone continuity (bony bridging) present in three out of four cortices in two projections (anterior-posterior & lateral x-rays), assessed by a blinded senior orthopedic surgeon.
  CT scan, for confirm the results

SECONDARY OUTCOMES:
Pain | 3months
  The pain relief as measured by Visual Analogue Scale (VAS) 3 months after cell injection
Quality of life | 3months
  Evaluation the patients' quality of life with Visual Analogue Score (VAS) 3months after cell transplantation.
Walking distance | 3months
  Walking distance changes as measured by walking on treadmill 3 months after cell injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Regenerative medicine department and cell therapy center of Royan Institute; Mohammad Razi, MD, Study Director — Department of orthopedic surgery, Tehran university of medical science, Tehran, Iran; Mohsen Emadedin, MD, Principal Investigator — Cell therapy center of Royan Institute; Narges Labibzadeh, MD, Principal Investigator — Department of Regenerative Medicine and cell therapy center, Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://RoyanInstitute.org